CLINICAL TRIAL: NCT01645371
Title: Assessing the Content Validity of a Stool Symptom Screener in Patients With Chronic Opioid-Induced Constipation
Brief Title: Assessing a Stool Symptom Screener in Patients With Chronic Opioid-Induced Constipation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3820C00028
Record Dates: First submitted 2012-07-12; First posted 2012-07-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Opioid-induced Constipation
Keywords: opioid-induced constipation
MeSH Terms: conditions — Opioid-Induced Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with opioid induced constipation

SUMMARY:
This qualitative research is to assess the validity of the stool symptom screener that will be used in patients with chronic opioid-induced constipation to determine the adequacy of their response to laxatives.

DETAILED DESCRIPTION:
Assessing the Content Validity of a Stool Symptom Screener in Patients with Chronic Opioid-Induced Constipation

ELIGIBILITY:
Inclusion Criteria:

* Receiving a stable maintenance opioid regimen (total daily dose of 30-1000mg of oral morphine, or equianalgesic amounts of 1 or more other opioid therapies) for a minimum of 4 weeks for non-cancer related pain.
* Development of constipation symptoms since starting opioids.
* Taken laxatives to help with bowel movements for at least four days over the past 2 weeks.

Exclusion Criteria:

* Receiving opioid regimen for treatment of pain related to cancer.
* Participated in any clinical trial or research study relating to opioid use and/or constipation within the past year.
* History of cancer within 5 years from the time of screening.
* Has medical condition(s) and/or treatment(s) associated with diarrhea, intermittent loose stools, or constipation (e.g., fecal incontinence or chronic idiopathic constipation).
* Has irritable bowel syndrome (IBS) or chronic functional constipation.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multi-speciality medical clinics ( family practice, neurology, internal medicine, pain management)
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Semi-structured discussion guide | Data will be collected at ONE time point from each patient using a semi-structured interview guide (up to 5 months)
  Using a semi-structured discussion guide during a single one-on-one interview, qualitative information will be collected from subjects that relates to their experience with Opioid Induced Constipation symptoms and to their understanding and perception of a verbally-administered stool symptom screener.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Karin S Coyne, PHD, MPH, Principal Investigator — United BioSource

REFERENCES:
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Slappendel R, Simpson K, Dubois D, Keininger DL. Validation of the PAC-SYM questionnaire for opioid-induced constipation in patients with chronic low back pain. Eur J Pain. 2006 Apr;10(3):209-17. doi: 10.1016/j.ejpain.2005.03.008. PMID 15914049
- See also: D3820C00028_statement_of_no_CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1400&filename=Study_D3820C00028_statement_of_no_CSR_Synopsis.pdf